CLINICAL TRIAL: NCT06642610
Title: CGM Dynamic Index (CDI) for Predicting Prediabetes in People With Cystic Fibrosis
Brief Title: CGM Dynamic Index for Predicting Prediabetes in Cystic Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Viral N. Shah, Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24262; DartCF funded by NIH/ NIDDK (Other Grant/Funding Number: Dartmouth Cystic Fibrosis Research Center (DartCF))
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Prediabetes; Cystic Fibrosis (CF); Cystic Fibrosis-related Diabetes
MeSH Terms: conditions — Prediabetic State; Cystic Fibrosis | interventions — Models, Theoretical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CF without diabetes (Other): a person with cystic fibrosis and no diabetes
  Interventions: Device: CGM Dynamic Index (CDI)
- CF with Prediabetes (Other): a person with cystic fibrosis and prediabetes
  Interventions: Device: CGM Dynamic Index (CDI)

INTERVENTIONS:
Device: CGM Dynamic Index (CDI) — Participants will undergo one-time oral glucose tolerance test (OGTT) and a one-time use of a CGM device, which will be worn for up to 10 days.
  Other Names: CGM Dynamic Index (CDI) mathematical model

SUMMARY:
The primary objective of this pilot study is to develop a CGM-based model to predict the progression from prediabetes to diabetes in individuals with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* CF individuals aged 12-55 years.
* CF without diabetes or with prediabetes (as defined by OGTT and HbA1c).
* Willing to use a continuous glucose monitoring system with compatible smart phone for glucose data collection.

A person with CFRD and already using CGM, we will just collect their personal CGM data, and they are not required to have OGTT or HbA1c visit.

Exclusion Criteria:

* Pregnancy.
* History of transplant.
* Use of immunosuppressant drugs.
* Use of oral steroids or any medication known to interfere with glucose.
* Allergy to adhesives.
* Individuals with severe concurrent medical conditions that could confound glucose monitoring data (e.g., terminal illness, major organ failure).
* Conditions that may make unsafe for participants to do study or impair or confound the study at the discretion of the investigator

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CGM Dynamic Index (CDI) for predicting prediabetes in people with cystic fibrosis | 10 days
  Estimating the "optimal" cut-offs of the CDI marker, to distinguish between CF groups

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health, University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided